CLINICAL TRIAL: NCT02221349
Title: A Randomized Clinical Study of the Safety and Effectiveness of Two Dentinal Hypersensitivity Treatments Used With Normal Oral Hygiene
Brief Title: A Clinical Study of Two Dentinal Hypersensitivity Treatments Used With Normal Oral Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014069
Record Dates: First submitted 2014-08-12; First posted 2014-08-20 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxalate liquid & gel plus SnF2 paste (Other): Potassium oxalate liquid, professionally applied Potassium oxalate gel, self applied Stannous fluoride paste, self applied
  Interventions: Device: Potassium oxalate; Drug: Stannous fluoride paste
- oxalate liquid & gel plus NaF paste (Other): Potassium oxalate liquid, professionally applied Potassium oxalate gel, self applied Sodium fluoride paste, self applied
  Interventions: Device: Potassium oxalate; Drug: Sodium fluoride paste

INTERVENTIONS:
Device: Potassium oxalate — Professionally applied (liquid) and self applied (gel)
Drug: Sodium fluoride paste — Toothpaste used by subject
  Other Names: NaF paste
  Arms: oxalate liquid & gel plus NaF paste
Drug: Stannous fluoride paste — Toothpaste used by subject
  Other Names: SnF2 paste
  Arms: oxalate liquid & gel plus SnF2 paste

SUMMARY:
This study will compare the safety and effectiveness of normal oral hygiene with two different marketed dentifrices, on longer term dentinal hypersensitivity response following use of potassium oxalate desensitizers.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written informed consent prior to participation and be given a signed copy of the informed consent form
* Complete a confidentiality disclosure agreement
* Be in good general health as determined by the Investigator/designee
* Have at least one tooth with a Schiff sensitivity score of at least 1 in response to the air challenge.

Exclusion Criteria:

* Self-reported pregnancy or nursing
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession
* Active treatment of periodontitis
* Fixed facial orthodontic appliances
* A history of kidney stones
* Known allergies to the following ingredients; aqua, glycerin, cellulose gum, dipotassium oxalate, carbomer, sodium hydroxide, sodium benzoate, and potassium sorbate
* Any diseases or conditions that might interfere with the safe completion of the study
* An inability to undergo any study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad J Anderson, MS, DMD, Principal Investigator — Chad J Anderson DMD Inc
Locations (1):
- Chad J Anderson DMD Inc, Fresno, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxalate Liquid & Gel Plus SnF2 Paste | Oxalate Liquid & Gel Plus NaF Paste
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxalate Liquid & Gel Plus SnF2 Paste | Oxalate Liquid & Gel Plus NaF Paste | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.97) | 44.9 (12.52) | 43.2 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1 | 2 | 3
  American Indian | 0 | 1 | 1
  Asian Oriental | 2 | 0 | 2
  Black | 2 | 0 | 2
  Caucasian | 10 | 11 | 21
  Multi-Racial | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows: 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subjects responds to stimulus and requests discontinuation or moves from stimulus, 3: tooth/subject responds to stimulus considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The mean change from Baseline was calculated for this measure.
Time Frame: 60 days
Population: Thirty (30) subjects received study products and were measured at the Baseline visit. Twenty-Nine (29) subjects completed the study thus, one subject dropped from the study prior to Day 60 and was not analyzed for the 60 day measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Liquid & Gel Plus SnF2 Paste | Oxalate Liquid & Gel Plus NaF Paste
Number analyzed (Participants) | 14 | 15
Units on a scale | -1.643 (0.770) | -1.500 (0.906)

2. Secondary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced.
Time Frame: 60 days
Population: Thirty (30) subjects received study products. Twenty-Nine (29) subjects completed the study thus, one subject dropped from the study prior to Day 60 and was not analyzed for the 60 day measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Liquid & Gel Plus SnF2 Paste | Oxalate Liquid & Gel Plus NaF Paste
Number analyzed (Participants) | 14 | 15
Units on a scale | -29.82 (18.65) | -24.67 (26.75)

ADVERSE EVENTS:
Arm/Group | Oxalate Liquid & Gel Plus SnF2 Paste | Oxalate Liquid & Gel Plus NaF Paste
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 1/14 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxalate Liquid & Gel Plus SnF2 Paste (N=14) | Oxalate Liquid & Gel Plus NaF Paste (N=15)
Hyperesthesia (Gastrointestinal disorders) | 1 (2) | 0 (0) — Burning and painful mouth
PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) — Painful mouth, mild and possibly related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes